CLINICAL TRIAL: NCT05639010
Title: A Multi-center, Open-label, Randomized Trial of Hemodialysis Plus Hemoperfusion on Blood β2-microglobulin (β2-MG), Parathyroid Hormone (PTH) and C Reactive Protein (CRP) Clearance in Maintenance Hemodialysis Patients
Brief Title: Effects of Hemodialysis Plus Hemoperfusion in Maintenance Hemodialysis Patients: A Clinical Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Changhai Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHEC2022-207
Record Dates: First submitted 2022-11-06; First posted 2022-12-06 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-06

CONDITIONS: End Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Renal Dialysis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- regular hemodialysis (Active Comparator): Routine blood purification therapy (including hemodialysis, hemofiltration) 3 times a week
  Interventions: Device: regular hemodialysis
- hemoperfusion combined with hemodialysis (Experimental): Routine blood purification therapy 3 times a week + Combination of hemodialysis and hemoperfusion treatment once a week
  Interventions: Device: regular hemodialysis; Device: hemoperfusion combined with hemodialysis

INTERVENTIONS:
Device: regular hemodialysis — Routine blood purification therapy (including hemodialysis, hemofiltration) 3 times a week
Device: hemoperfusion combined with hemodialysis — Hemoperfusion combined with hemodialysis treatment will perform once a week. The hemoperfusion apparatus will use type KHA80 hemoperfusion apparatus (Zhuhai Jafron Biomedical Co., Ltd, China)
  Arms: hemoperfusion combined with hemodialysis

SUMMARY:
This multi-center, open-label, randomized, parallel controlled trial aims to investigate the efficacy of hemoperfusion (HP) in combination with hemodialysis (HD) by assessing blood β2-microglobulin (β2-MG), parathyroid hormone (PTH) and C reactive protein (CRP) clearance in maintenance hemodialysis patients.

DETAILED DESCRIPTION:
In this HD/HP vs HD trial, the investigators plan to enroll 410 maintenance hemodialysis patients. Twelve medical centers in the Shanghai metropolitan area have expressed interest in participating. Participants will be randomized into 2 groups after a 1-month washout period. The control group (205 patients) will be treated with hemodialysis or hemofiltration with a frequency of 3 times/week; the experimental group (205 patients) will be treated with Jafron KHA80 hemoperfusion apparatus in addition to hemodialysis or hemofiltration with a frequency of 1 time/week. Follow-up data before the last dialysis at 4, 12, 24, 36 and 52 weeks of treatment were collected from both groups, including the following: routine physical examination, laboratory tests (blood routine, blood biochemistry, β2-MG, PTH, CRP, liver/kidney function, coagulation system tests, etc.), chest X-ray, electrocardiogram and cardiac ultrasound. Dialysis adequacy as defined by standard Kt/V will be calculated. Comorbidities, combined medications and adverse events will also be captured. The primary outcomes will include change in blood β2-MG, PTH and CRP values. Secondary outcomes will include change values for serum protein-bound toxins (e.g., p-Cresol sulfate, indophenol sulphate), improvement in patient quality of life (Kidney Disease Quality of Life Short Form), sleep disturbance (Pittsburgh Sleep Quality Index) and pruritus (Duo's pruritus score).

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80 years, regardless of gender
2. Stable maintenance hemodialysis for ≥ 3 months with relatively fixed dialysis pattern
3. Hemodialysis treatment 3 times per week, total treatment duration ≥ 10 hours per week, vascular access unlimited
4. Blood β2-MG > 30 mg/L and/or 300 pg/ml < immunoreactive parathyroid hormone (iPTH) < 800 pg/ml and/or CRP ≥ 16.2 pg/ml
5. Kt/V ≥ 1.2 eight weeks prior to enrollment
6. Signed informed consent form

Exclusion Criteria:

1. Known allergic reaction, contraindication or intolerance to the material of the dialyzer or perfusion apparatus
2. Test indicators meeting one or more of the following: white blood cell <4 x 10^9/L, platelet count <60 x 10^9/L, serum albumin <30 g/L
3. Blood flow <200 ml/min
4. Regular hemoperfusion treatment for more than 3 months and at least once every 2 weeks
5. Active bleeding or chronic gastrointestinal bleeding, or other severe bleeding tendencies or coagulation disorders
6. History of unstable angina pectoris, myocardial infarction, severe arrhythmia, pericarditis, myocarditis, cardiac surgery or peripheral vascular surgery in the last 8 weeks
7. Cerebral hemorrhage in the last 12 weeks
8. Severe heart failure (New York Heart Association class IV)
9. Acute infection, acute or critical illnesses such as severe cardiac, pulmonary, hepatic or neurological disease and malignancy
10. Pregnancy or breastfeeding
11. Participation in a clinical trial or ongoing clinical trial within 3 months
12. Expected survival of less than 1 year
13. Not considered suitable for participation in this trial by the investigator

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 410 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in blood β2-microglobulin (β2-MG) values | From date of enrollment until the end of study, assessed up to 52 weeks
  Compared the difference between standardized therapy and hemoperfusion combined with hemodialysis treatment on the clearance of blood β2-MG in maintenance hemodialysis patients
Changes in blood Parathyroid Hormone (PTH) values | From date of enrollment until the end of study, assessed up to 52 weeks
  Compared the difference between standardized therapy and hemoperfusion combined with hemodialysis treatment on the clearance of blood PTH in maintenance hemodialysis patients
Changes in blood C Reactive Protein (CRP) values | From date of enrollment until the end of study, assessed up to 52 weeks
  Compared the difference between standardized therapy and hemoperfusion combined with hemodialysis treatment on the clearance of blood CRP in maintenance hemodialysis patients

SECONDARY OUTCOMES:
Change in serum protein-bound toxin (e.g., p-Cresol sulfate, indophenol sulphate) values | From date of enrollment until the end of study, assessed up to 52 weeks
  Compared the difference between standardized therapy and hemoperfusion combined with hemodialysis treatment on the clearance of serum protein-bound toxin (e.g., p-Cresol sulfate, indophenol sulphate) in maintenance hemodialysis patients
Improvement in patients' quality of life | From date of enrollment until the end of study, assessed up to 52 weeks
  Assessment of quality of life using the Kidney Disease Quality of Life Short Form (KDQOL-SF) questionnaire
Improvement in patients' sleep disturbance | From date of enrollment until the end of study, assessed up to 52 weeks
  Assessment of sleep disturbance using the Pittsburgh Sleep Quality Index (PSQI)
Improvement in patients' pruritus | From date of enrollment until the end of study, assessed up to 52 weeks
  Assessment of pruritus using the Duo's pruritus score

CONTACTS AND LOCATIONS:
Overall Officials: Zhiyong Guo, professor, Study Director — Changhai Hospital
Locations (1):
- Changhai Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the publication article, after deidentification (text, tables, figures, and appendices), will be shared.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The available data period begins 3 months and ends 5 years following the article's publication.
Access Criteria: Investigators who provide a methodologically sound proposal for scientific research with non-commercial purposes will be able to access the IPD and supporting information.
  Deidentified participant data that underlie the results reported in the publication article will be shared, which can be available from Professor Zhiyong Guo (contacting email: drguozhiyong@163.com, ORCID: Shenneike66). Proposals should be directed to drguozhiyong@163.com. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Derived] Huang W, Zhang L, Wu H, Chen W, Guo Z. Effects of combined haemodialysis-haemoadsorption therapy in maintenance haemodialysis patients: study protocol for a multicentre, open-label, randomised, parallel controlled trial. BMJ Open. 2025 Nov 12;15(11):e107017. doi: 10.1136/bmjopen-2025-107017. PMID 41224301